CLINICAL TRIAL: NCT04026100
Title: A Phase I Clinical Trial of CTA101 UCART Cells Injection in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: CTA101 in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-CTA101
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTA101 (Experimental)
  Interventions: Biological: CTA101

INTERVENTIONS:
Biological: CTA101 — Universal CD19-directed CAR-T cells by a single infusion intravenously will be given in escalating doses. Subjects will been distributed into low dose (0.2×10^6), medium dose (2×10^6), and high dose (3×10^6).

SUMMARY:
This is a single-center, non-randomized and dose-escalation study to evaluate the safety and efficacy of CTA101 in relapsed or refractory diffuse large B-cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of DLBCL per WHO Classification Criteria for Lymphocytic Tumors 2016, including DLBCL and PMBCL transformed from follicular lymphoma;
2. Relapsed or refractory DLBCL (meeting one of the following conditions):

   1. Recurrence, progression or stable disease (SD) after treatment with second-line or above second-line chemotherapy regimens;
   2. Recurrence or progression after autologous hematopoietic stem cell transplantation;
3. At least one measurable lesion must be ≥ 1.5cm in the longest diameter;
4. Male or female aged 18-70 years;
5. Estimated survival time ≥ 12 weeks;
6. Serum albumin ≥ 30g/L, total bilirubin ≤ 25.7umol/L, creatinine ≤ 132.6umol/L, alanine transaminase (ALT) and aspartate aminotransferase (AST) <3 times of upper limit of normal;
7. Absolute neutrophil count ≥ 1.0*10^9/L, platelet count ≥ 50*10^9/L;
8. ECOG performance status 0 to 1;
9. Echocardiographic diagnosis shows left ventricular ejection fraction (LVEF) ≥ 50%;
10. No active infection in the lungs;
11. Latest treatment (radiotherapy, chemotherapy, monoclonal antibody therapy or other treatment) must have been completed at least 2 weeks prior to screening;
12. All women of child-bearing potential must have a negative blood or urine pregnancy test at screening, and agree to take medically acceptable contraception measures while on study treatment;
13. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. History of hypersensitivity to any component of cell product;
2. Prior treatment with any CAR T cell product or other genetically-modified T cell therapies;
3. Recurrence after allogeneic hematopoietic stem cell transplantation;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis), or currently receiving antibiotic therapy by intravenous drip. However, prophylactic antibiotic, antiviral and antifungal treatments are allowed;
5. HBV DNA copy number detected by PCR in patients with active hepatitis B is > 1000 at screening (if HBsAg positive, routine antiviral therapy is required after enrollment), as well as CMV, hepatitis C, syphilis and HIV infection;
6. Patients with New York Heart Associate (NYHA) Class III/IV cardiac insufficiency (see Appendix 1);
7. Patients with Corrected QT interval(QTc)>450 msecs (Fridericia formula);
8. Patients with a history of epilepsy;
9. Intracranial extranodal lesions (tumor cells in cerebrospinal fluid, and/or MRI shows intracranial lymphoma invasion);
10. Extensive invasions of gastrointestinal lymphoma (lesions involving the muscular layer, serosa and subserosa, excluding lesions confined to the mucosa and submucosa);
11. History of other primary cancer, except for the following conditions:

    1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin
    2. Cured carcinoma in situ, such as cervical cancer, bladder cancer or breast cancer
12. Patients with autoimmune diseases requiring treatment, patients with immunodeficiency or requiring immunosuppressive therapy;
13. Concurrent therapy with systemic steroids within 1 week prior to screening, except for the patients recently or currently receiving inhaled steroids;
14. Women pregnant or lactating, with a pregnancy plan within 6 months, fertile but unable to take medically acceptable contraception measures;
15. Patients who have participated in any other clinical studies within 2 weeks prior to screening;
16. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | Baseline up to 35 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v4.03 criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) | 4 weeks, 12 weeks, 6 months, 12 months, 18 months and 24 months
  Assessment of overall response rate for weeks 4, 12, months 6, 12, 18 and 24 in accordance with Lugano 2014 (overall response rate，OR)
Disease control rate (DCR) | 12 weeks, 6 months, 12 months, 18 months and 24 months
  Assessment of overall response rate for weeks 12, months 6, 12, 18 and 24 in accordance with Lugano 2014（disease control rate，DCR)

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China